CLINICAL TRIAL: NCT03570736
Title: Evaluation of Gain In Clinical Attachment And Bone Levels After Treatment of Patients With Intra-bony Defects By Minimally Invasive Surgical Technique Versus Open Flap Debridement. A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Gain In Clinical Attachment And Bone Levels After Treatment of Patients With Intra-bony Defects By Minimally Invasive Surgical Technique Versus Open Flap Debridement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal El Din Abd El Salam, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12348765
Record Dates: First submitted 2018-06-14; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Minimally Invasive Surgical Technique; Open Flap Debridement; Microsurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Invasive Surgical Technique (Experimental)
  Interventions: Procedure: Minimal invasive surgical technique
- Open Flap Debridement (Active Comparator)
  Interventions: Procedure: Open Flap Debridement

INTERVENTIONS:
Procedure: Minimal invasive surgical technique — Minimal Invasive Surgical technique using either Modified Papilla Preservation or Simplified Papilla Preservation Technique.
  Arms: Minimal Invasive Surgical Technique
Procedure: Open Flap Debridement — Buccal and lingual intrasulcular incisions will be done extending at least one tooth mesial and distal to the tooth associated with the intrabony defect. Full thickness mucoperiosteal flaps will be reflected to allow access for debridement of the defect.
  Arms: Open Flap Debridement

SUMMARY:
Hypothesis:The conventional surgical approach is to raise large flaps to completely and exceedingly expose the area of interest. Since the results were unsatisfactory due to limited regenerated periodontal tissue, an alternative approach to access the intra-bony defects was proposed, this approach is called minimally invasive techniques which use incisions just large enough for debridement and generally involves reflecting the papilla only using specialized instruments to access the intra-bony defect and debridement.

Aim of the study:Is to evaluate the gain in clinical attachment level and bone after treatment of the intra-bony defects by Minimally Invasive Surgical Technique when compared to Open Flap Debridement in patients with intra-bony defects.

Study setting:Study will be conducted in the Oral Medicine and Periodontology department, Faculty of Oral and Dental Medicine - Cairo University, Egypt.Patients will be selected from the outpatient clinic of the department of Oral Medicine and Periodontology-Cairo University.

Prior to the start of the study each patient will receive initial periodontal therapy consisting of proper oral hygiene instructions and full-mouth scaling and root planing. Six weeks after completion of the initial therapy, a re-evaluation will be performed to confirm that the patients meet all the inclusion criteria for the study.

Evaluation of the patient's oral hygiene and a written consent will be obtained from the patients who will participate in the trial. Blinded periodontist will record the clinical measurements prior to surgery using a periodontal probe.

Prior to surgery, a stent will be fabricated for each site using diagnostic casts and acrylic resin. Each stent will rest on the occlusal surfaces of at least 4 teeth and had a vertical notch marking the facial and lingual position of the intra-bony defect. A periapical radiograph using paralleling technique using extension cone paralleling (XCP) film holder will be performed for each patient to evaluate alveolar bone loss using DIGORA system.

Surgical procedure:The patients will be randomly assigned into two groups; Group A (Control): Patients receiving Open Flap Debridement (OFD). Group B (Test): Patients receiving Minimally Invasive Surgical technique (MIST).

The operator will anesthetize the surgical sites for both groups. For the OFD technique, buccal and lingual intrasulcular incisions will be done extending at least one tooth mesial and distal to the tooth associated with the intrabony defect. Full thickness mucoperiosteal flaps will be reflected to allow access for debridement of the defect.

Surgical debridement will be carried out to remove subgingival plaque, calculus and granulation tissue. The surgical sites will be irrigated with sterile saline. Surgical flaps will be sutured to the pre-surgical level with 5-0 vicryl suture utilizing a vertical mattress suturing technique achieving primary closure.

For the Minimally Invasive Surgical technique, it will be carried out with 2.5 X optical magnification dental loupes. After local anaesthesia, an envelope flap without vertical releasing incisions will be performed. The defect-associated interdental papilla will be accessed either with the simplified papilla preservation flap (SPPF) in narrow interdental spaces or the modified papilla preservation technique (MPPT) in large interdental spaces. In the SPPF, a diagonal incision traced as close as possible to the buccal side of the papilla col will be performed, whereas in the MPPT a horizontal incision traced on the buccal side of the papilla will be done. Intrasulcular incisions will be performed from the interdental side to the buccal and lingual sides of the teeth neighboring the defect; tiny buccal and lingual flaps will be elevated to expose the bone crest.

All incisions will be done using microsurgical ophthalmic blades. Buccal and lingual flaps will be elevated using sharp dissection only. Granulation tissue adherent to the inner surface of flaps will be carefully removed with microscissors to provide full access and visibility to root surfaces. Defect debridement and root planing will be performed with a combination of mini-curettes. Then sutures will be placed using 6-0 vicryl suture.

Postoperative medication:Administration of amoxicillin (500 mg tabs) T.I.D for 7 days), Chlorhexidine rinse (B.I.D for 14 days). Ibuprofen 600 mg tabs 1 every 8h in case of unbearable pain.

Patient self-care instructions: Sutures will be removed 2 weeks post-surgically. Patients will be asked to abstain from mechanical oral hygiene procedures in the surgical area for 2 weeks. After this period, patients will be instructed to continue mechanical tooth brushing again of the treated sites using a soft toothbrush.

The outcomes will be measured at 1 week, 3 and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* 25 years of age or older.
* At least one periodontal infrabony pocket (detected radiographically) with Probing depth (PD) ≥5 mm,
* Plaque index < 30 %

Exclusion Criteria:

* Hopeless tooth.
* Previous periodontal surgery within the last 2 years in area of interest.
* Systemic conditions which are generally considered to be a contraindication to periodontal surgery which included but not limited to: osteoporosis, uncontrolled diabetes.
* Pregnant or lactating females
* Current or former smokers.
* Non compliant patients

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | up to 6 months post-operatively
  It is the distance measured from the cemento-enamel junction (CEJ) to the bottom of the pocket.

SECONDARY OUTCOMES:
Probing Depth | up to 6 months post-operatively
  It is the distance measured from the gingival margin to the bottom of the pocket.
Gingival Recession | up to 6 months post-operatively
  It is the distance measured from the CEJ to the most apical extension of gingival margin.
Post-Operative Pain | up to 1 week post-operatively
  It wil be measured by Visual Analogue Scale (VAS) with numbers from 0 to 10 (0 indicates 'no pain' to 10 which indicates 'worst pain imaginable')
Bone Fill | up to 6 months post-operatively
  It will be measured radio-graphically by DIGORA system

IPD SHARING:
Plan to Share IPD: Undecided